CLINICAL TRIAL: NCT04600258
Title: Chocolate for the Patient With Chronic Kidney Disease: a New Strategy to Modulate Inflammation?
Brief Title: Chocolate for Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Denise Mafra, Full Professor, Universidade Federal Fluminense
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: DeniseMafra10
Record Dates: First submitted 2020-10-18; First posted 2020-10-23 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Chocolate group Control Group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chocolate Group (Experimental): Administration of 40g dark chocolate per day, for 2 months
  Interventions: Dietary Supplement: Dark Chocolate
- Control Group (No Intervention): No intervention and analysis will be performed before and after 2 months

INTERVENTIONS:
Dietary Supplement: Dark Chocolate — The patients will receive 40g per day of dark chocolate for 2 months
  Arms: Chocolate Group

SUMMARY:
Chocolate is a widely appreciated foodstuff with historical appreciation as food from the gods. It is a rich source of (poly)phenolics, which have several proposed salutogenic effects, including neuroprotective anti-inflammatory, antioxidant, and cardioprotective properties.

This study will evaluate the potential salutogenic contribution of chocolate intake, to mitigate inflammatory and oxidative burden in chronic kidney disease patients.

DETAILED DESCRIPTION:
This study is evaluating patients with CKD on a regular HD program randomized in the chocolate group and control group. The chocolate group is receiving 40g of dark chocolate per day for 2 months and the control group is not receiving any intervention. Peripheral blood mononuclear cells (PBMC) are being isolated for expression of Nrf2, NF-kB, and NADPH quinone oxidoreductase 1 (NQO1) by a quantitative real-time polymerase chain reaction. Antioxidant enzymes activity (catalase-CAT and glutathione peroxidase-GPx), high-sensitivity C-reactive protein (hs-CRP) will be assessed using an enzyme-linked immunosorbent assay (ELISA).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Chronic Kidney Disease
* Hemodialysis patients for more than 6 months
* Aged 18 years or older

Exclusion Criteria:

* Patients pregnant
* Smokers
* Using antibiotics in the last 3 months
* Autoimmune diseases
* Clinical diagnosis of infectious diseases
* Clinical diagnosis of Cancer
* Clinical diagnosis of AIDS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Antioxidants and anti-inflammatory biomarkers | 2 months
  Get blood samples to evaluate the supplementation effects in antioxidants biomarkers- nuclear receptor factor 2 (Nrf2), glutathioneperoxidase (GPx), heme oxygenase-1 (HO-1)
Inflammatory biomarkers | 2 months
  Get blood samples to evaluate the supplementation effects in inflammatory biomarkers- factor nuclear kappa B (NFkB), interleukin 6 (IL-6), tumor necrosis factor alpha (TNF-alpha)

SECONDARY OUTCOMES:
Uremic toxins | 2 months
  Get blood samples to evaluate the supplementation effects on uremic toxins plasma levels

CONTACTS AND LOCATIONS:
Locations (1):
- Denise Mafra, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fanton S, Cardozo LFMF, Combet E, Shiels PG, Stenvinkel P, Vieira IO, Narciso HR, Schmitz J, Mafra D. The sweet side of dark chocolate for chronic kidney disease patients. Clin Nutr. 2021 Jan;40(1):15-26. doi: 10.1016/j.clnu.2020.06.039. Epub 2020 Jul 14. PMID 32718711
- [Derived] Kemp JA, Fanton S, Baptista BG, Ribeiro M, Cardozo LFMF, Ribeiro-Alves M, Mafra D. Short Report: Influence of Dark Chocolate Intake on Magnesium Status in Hemodialysis Patients. J Ren Nutr. 2025 Jul;35(4):545-549. doi: 10.1053/j.jrn.2025.02.002. Epub 2025 Feb 26. PMID 40020766
- [Derived] Kemp JA, Schultz J, Modolon F, Ribeiro-Alves M, Rosado AS, Mafra D. Is there a correlation between TMAO plasma levels and archaea in the gut of patients undergoing hemodialysis? Int Urol Nephrol. 2025 Apr;57(4):1269-1275. doi: 10.1007/s11255-024-04273-5. Epub 2024 Nov 19. PMID 39562414
- [Derived] Ribeiro M, Fanton S, Paiva BR, Baptista BG, Alvarenga L, Ribeiro-Alves M, Cardozo LF, Mafra D. Dark chocolate (70% cocoa) attenuates the inflammatory marker TNF-alpha in patients on hemodialysis. Clin Nutr ESPEN. 2023 Feb;53:189-195. doi: 10.1016/j.clnesp.2022.12.009. Epub 2022 Dec 9. PMID 36657913